CLINICAL TRIAL: NCT07311031
Title: Effect of Blood Flow Restriction Training on Quadriceps Muscle Strength, Knee Biomechanics and Rehabilitation After Anterior Cruciate Ligament Reconstruction in Active Workers
Brief Title: Effect of Blood Flow Restriction Rraining on Rehabilitation After Anterior Cruciate Ligament Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital MAZ (Other)
Responsible Party: Principal Investigator, Raul Zapata Rodrigo, Orthopaedic Surgeon, Hospital MAZ
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAZ Hospital
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation; Blood Flow Restriction (BFR) Training Effects
Keywords: KAATSU; Knee injury; ACL rehabilitation
MeSH Terms: conditions — Knee Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFRT rehabilitation group (Experimental): Receive standard ACL physical therapy plus blood flow restriction training
  Interventions: Other: Blood flow restriction training; Other: Standard ACL rehabilitation
- Standard rehabilitation group (Active Comparator): Receive standard ACL physical therapy
  Interventions: Other: Standard ACL rehabilitation

INTERVENTIONS:
Other: Blood flow restriction training — BFRT consists of a pressurized cuff that is applied to the proximal thigh in order to partially occlude blood flow while the patient exercises. It is believed that the accumulated effects of fatigue, mechanical tension, metabolic stress and reactive hyperaemia contribute to promoting adaptation of the quadriceps with minimal strain. Therefore, patients can train at reduced loads and may receive the same training benefits as if they were training with high loads.
  Arms: BFRT rehabilitation group
Other: Standard ACL rehabilitation — A 14-16-week supervised accelerated early rehabilitation protocol was selected based on previous evidence.8 It is characterised by early unrestricted motion and weight-bearing, without the use of an immobilising brace and commencing early strength training.

SUMMARY:
Importance: Following anterior cruciate ligament reconstruction (ACLR), patients often experience quadriceps muscle weakness and atrophy, frequently leading to long-term complications. A promising rehabilitation program based on blood flow restriction training (BFRT) seems to be particularly valuable for patients who may be unable to train with heavy loads due recent surgery. Previous studies have demonstrated that BFRT promotes strength gains and muscle mass increases, with adaptations comparable to traditional high-intensity training, despite using low-load resistance exercises.

Objective: to evaluate the effect of blood flow restriction training on quadriceps strength and knee biomechanics in a 4-month rehabilitation program of patients who have had an ACL reconstruction.

Design: The study will be a two-arm superiority randomized controlled clinical trial.

Setting: The trial will be conducted at a work-related injuries specialised hospital, MAZ Hospital, Zaragoza, Spain.

Participants: Participants will be active workers who have suffered an acute ACL tear and they have undergone ACL reconstruction (n=60).

Intervention: Patients will recieve a 14-16-week supervised accelerated early rehabilitation protocol; one group will complete it applying blood flow restriction training and the other will not.

Main Outcome and Measure: The primary outcomes will be peak quadriceps strength and rate of torque development measured both isometrically and isokinetcally with a Isokinetic Dynamometer CON-TREX MG.

Limitations: Potential limitations include patients and physiotherapists are not blinded.

Conclusions: The focus of the research will examine the impact of blood flow restriction rehabilitation on patients who have undergone ACLR.

Relevance: The study has potential to restore quadriceps strength to a greater extent than standard rehabilitation protocol. Moreover, patients will spend less time in the rehabilitation process to return to work compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (18-65 years of age); must be skeletally mature with closed physes
* Worker active
* Diagnosis of acute (<8 weeks), unilateral ACL tear with planned surgery confirmed via clinical examination and MRI
* No previous ACL injury or reconstruction on the involved limb
* Planned graft: autologous ipsilateral hamstring graft for ACL reconstruction
* Planned fixation: suspensory cortical femoral device and tibial interference screw

Exclusion Criteria:

* Completed knee dislocation or multiligament injury (PCL, MCL, LCL)
* ACL Graft diameter < 8mm
* Meniscal suture or meniscal root reattachment
* Post-surgical immobilization
* Any current or previous conditions or surgeries that might affect gait
* Pregnant
* Spinal fusion
* Any implanted medical device or other contraindications for MRI
* History of deep vein thrombosis and/or varicose veins or familiy history of deep vein thrombosis
* Taking anti-coagulant drugs for any blood, cardiac or congenital disease that may cause coagulation disorders
* Taking bone and muscle metabolism-modulation drugs or muscle supplements (e.g., creatine, amino acids, whey protein,…)
* Recent inflammation, bleeding disorders, active bleeding, or infection within the lower limbs
* Diabetic or have uncontrolled hypertension
* Diminished capacity to provide informed consent
* Unfeasible to attend regular physical therapy and study visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Quadriceps strength | From enrollment to the end of treatment at 14 weeks
  Peak quadriceps strength
Quadriceps strength | From enrollment to the end of treatment at 14 weeks
  Rate of torque

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Casajus Mallen, University professor, Study Chair — Universidad de Zaragoza
Locations (1):
- MAZ Hospital, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Trained researchers will collect data from MAZ Hospital. All information collected during this trial will always be protected and securely stored by the lead researcher. The lead researcher will assign a secure locker in his office to store all investigation documents. Additionally, all electronic material will be safely stored and backed up on the researcher's computer equipment with a secure password.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Erickson LN, Lucas KCH, Davis KA, Jacobs CA, Thompson KL, Hardy PA, Andersen AH, Fry CS, Noehren BW. Effect of Blood Flow Restriction Training on Quadriceps Muscle Strength, Morphology, Physiology, and Knee Biomechanics Before and After Anterior Cruciate Ligament Reconstruction: Protocol for a Randomized Clinical Trial. Phys Ther. 2019 Aug 1;99(8):1010-1019. doi: 10.1093/ptj/pzz062. PMID 30951598
- [Background] Gopinatth V, Garcia JR, Reid IK, Knapik DM, Verma NN, Chahla J. Blood Flow Restriction Enhances Recovery After Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2025 Apr;41(4):1048-1060. doi: 10.1016/j.arthro.2024.05.032. Epub 2024 Jun 16. PMID 38889851
- [Background] Erickson LN, Owen MK, Casadonte KR, Janatova T, Lucas K, Spencer K, Brightwell BD, Graham MC, White MS, Thomas NT, Latham CM, Jacobs CA, Conley CE, Thompson KL, Johnson DL, Hardy PA, Fry CS, Noehren B. The Efficacy of Blood Flow Restriction Training to Improve Quadriceps Muscle Function after Anterior Cruciate Ligament Reconstruction. Med Sci Sports Exerc. 2025 Feb 1;57(2):227-237. doi: 10.1249/MSS.0000000000003573. Epub 2024 Oct 1. PMID 39350350
- [Background] Mather RC 3rd, Koenig L, Kocher MS, Dall TM, Gallo P, Scott DJ, Bach BR Jr, Spindler KP; MOON Knee Group. Societal and economic impact of anterior cruciate ligament tears. J Bone Joint Surg Am. 2013 Oct 2;95(19):1751-9. doi: 10.2106/JBJS.L.01705. PMID 24088967
- [Background] Matar HE, Platt SR, Bloch BV, James PJ, Cameron HU. A Systematic Review of Randomized Controlled Trials in Anterior Cruciate Ligament Reconstruction: Standard Techniques Are Comparable (299 Trials With 25,816 Patients). Arthrosc Sports Med Rehabil. 2021 May 14;3(4):e1211-e1226. doi: 10.1016/j.asmr.2021.03.017. eCollection 2021 Aug. PMID 34430902